CLINICAL TRIAL: NCT03040908
Title: Evaluation de la capacité Physique Sous Maximale au Moyen du Test de Marche de 6 Minutes Des Enfants et Adultes Jeunes Suivis Pour drépanocytose et Nouveaux paramètres d'hémolyse : Vers Une prédiction Des Complications Vasculaires ?
Brief Title: New Hemolysis Parameters in Sickle Cell Disease
Acronym: HEMODREP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2016/ONCO-HEMATO/HEMODREP
Record Dates: First submitted 2017-01-24; First posted 2017-02-02 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The 6-minute walk (6MWT) test is used in adults and children affected by a wide range of chronic diseases to evaluate their sub-maximal exercise capacity. It reflects the global response of various physiological systems (respiratory, cardio-vascular, neurologic, metabolic and musculosquelettic) in a situation simulating a daily life activity. In children with sickle cell disease, the 6MWT is correlated with a low level of hemoglobin, a low level of fetal hemoglobin and low red cell deformability. Our team previously reported that in a population of children with sickle cell disease, highly treated with hydroxyurea, the sole factor which was independently linked to the 6MWT was the presence of silence infarct.

As the cardio-vascular and cerebro-vascular injury in sickle cell disease are directly correlated with hemolysis, the investigators aim to evaluate a) the clinical relevance of endothelial and inflammation parameters and new hemolysis markers and b) if the presence of silent infarct and the 6MWT are correlated with this biological markers.

This cross-sectional study will include sickle cell disease patients regularly followed for more than 5 years at Hôpital Universitaire des Enfants Reine Fabiola, Centre Hospitalier Universitaire (CHU)-Brugmann, Centre Hospitalier Etterbeek-Ixelles, CHU Saint-Pierre, Cliniques Universitaires Saint-Luc (Bruxelles, Belgium). Inclusion criteria are: sickle cell disease (SS, Sbeta°, SC, Sbeta+), age range : 6 to 25 years, signed informed consent. Exclusion criteria are: transplanted patients, inability to perform the 6MWT (severe cognitive disability, femoral osteonecrosis with functional impairment), hospitalization and/ or transfusion in the last 3 months for acute event.

Demographic data and clinical data will be retrospectively recorded. Blood test and 6MWT will be performed in steady state. Studied analysis will be: coagulation factors, free hemoglobin, Pro-B type natriuretic peptide (Pro-BNP), High sensitivity C reactive protein (HS-CRP), Intercellular Adhesion Molecule (ICAM), Vascular Cell Adhesion Molecule (VCAM) and Selectins.

With this study, the investigators expect to validate new predictive markers for cardio-vascular or cerebrovascular injury and to identify patients at high risk to develop these complications.

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease (HbSS, S beta°, S beta+, SC)
* Regular follow-up from more than 5 years
* Written informed consent

Exclusion Criteria:

* Transplanted patients
* Hospitalisation for an acute event within 3 months
* Acute transfusion within 3 months
* Unable to performed 6-minute walk test

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults with Sickle Cell Disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between new biological data and clinical phenotype | 2 years
  The primary outcome of this study is to validate the relationship between these new biological markers and the clinical phenotype.

SECONDARY OUTCOMES:
Correlation between new biological data and 6-minute walk test | 2 years
  The secondary outcome is to confirm the correlation between the 6-minute walk test and the presence of silent infarct and to explore the relationship between these new markers and the 6-minute walk test.

IPD SHARING:
Plan to Share IPD: Undecided